CLINICAL TRIAL: NCT02927470
Title: Transcranial Magnetic Stimulation of Visual Working Memory
Brief Title: TMS of Visual Working Memory
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators are no longer at NYU Langone Health
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00666
Record Dates: First submitted 2016-10-04; First posted 2016-10-07 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Occipital Transcranial Magnetic Stimulation
Keywords: Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Working memory task (Experimental): Simple visual stimuli (e.g., dots, colors, lines) will be presented on a computer monitor. The positions of the stimuli must be attended and remembered and decisions about the stimuli and/or their locations must be made. Memory will be probed with a button press or an eye movement towards the remembered locations.
  Interventions: Device: Sham TMS condition; Device: OffLine TMS Condition; Device: Online TMS condition

INTERVENTIONS:
Device: Sham TMS condition — A sham TMS coil will be used to measure baseline performance on the working memory task. The sham coil looks and sounds just like the real coil, but produces a negligible magnetic field. Following the 40 seconds of sham TBS, the subject will perform the working memory task for 45 minutes.
Device: OffLine TMS Condition — A total of 200 trains will be delivered successively in 40 s, totaling 600 pulses. The pulses will be delivered at 80% of motor thresholds. A sham TMS coil will be used to measure baseline performance on the working memory task. The sham coil looks and sounds just like the real coil, but produces a negligible magnetic field. Following the 40 seconds of TBS, or sham TBS, the subject will perform the working memory task for 45 minutes.
Device: Online TMS condition — A single train of pulses (3 pulses at 50Hz, duration 40ms) will be delivered once during a particular time epoch on each trial, followed by a minimum of 6 seconds of no stimulation. No more than 600 pulses will be applied in a single session. Similar to the offline TMS condition, a sham TMS coil will be used to measure baseline performance on the working memory task. In each session (frontal, sham) subjects will perform the working memory task for 45 minutes.

SUMMARY:
The purpose of this study is to understand how the brain allows individuals to keep information "in mind" over brief intervals. During the experiment, participants will be asked to maintain fixation while they attend to and remember different visual stimuli (e.g., the location of a dot on the screen, the color of a circle, the orientation of a line, the speed of a group of moving dots) on a computer monitor. Participants will make decisions about these visual stimuli and indicate their decisions by pressing buttons or making eye movements. Through the use of Transcranial Magnetic Stimulation (TMS) investigators hope to understand the contributions of different anatomical areas while subjects perform this task.

DETAILED DESCRIPTION:
This study will use a within subject design in which each participant will perform a working memory task combined with Transcranial Magnetic Stimulation. TMS will be applied in three possible procedures, 1) Online TMS, 2) Offline TMS and 3) Sham TMS. All subjects will be given two trials within their one session, one of which will be sham TMS for all subjects and another of which will be randomly assigned to either Online or Offline TMS. Trials order will be randomly counterbalanced across subjects, who will be blind to the treatment of frontal vs. sham TMS (independent variable). Participants will be randomized into either the online or offline groups by computer generated lists to ensure equal numbers of participants in each condition. Half of the subjects will receive online TMS (online group) and half will receive offline TMS (offline group). Subjects will be randomly assigned to one of the two groups. The dependent variables will be performance accuracy and reaction time on the working memory task. By utilizing online and offline TMS, investigators will be able to explore whether frontal cortex is involved transiently in visual working memory or persistently throughout the task.

ELIGIBILITY:
Inclusion Criteria:

* Neurologically healthy individuals will be recruited.

Exclusion Criteria:

* Individuals with neurological issues (e.g., history of seizures, neurosurgery, brain trauma) will be excluded.
* Women of childbearing potential will be told that although there are no known risks of the procedure to the unborn fetus, they should not take part in the study if they are or might be pregnant.
* Minors and the elderly will be excluded.
* Individuals who are on medications that heighten the risk of TMS adverse events will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Performance Accuracy (number of correct button presses) on the working memory task | 1 Hour
  Simple visual stimuli (e.g., dots, colors, lines) will be presented on a computer monitor. The positions of the stimuli must be attended and remembered and decisions about the stimuli and/or their locations must be made. Memory will be probed with a button press or an eye movement towards the remembered locations.
Length of reaction time used in answering questions | 1 Hour
  Simple visual stimuli (e.g., dots, colors, lines) will be presented on a computer monitor. The positions of the stimuli must be attended and remembered and decisions about the stimuli and/or their locations must be made. Memory will be probed with a button press or an eye movement towards the remembered locations.

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sreenivasan, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States